CLINICAL TRIAL: NCT06546709
Title: A Phase 1, Randomized, Recipient- and Observer-Blinded, Dose-Escalation Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Two Doses of Rabies-Vectored Monovalent Lassa Fever Vaccine (LASSARAB) Administered With 3D-(6-Acyl) PHAD-SE (aPHAD-SE) Adjuvant in Healthy Adults
Brief Title: DMID 23-0015; Lassa Fever CVD 1000
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wilbur Chen, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Wilbur Chen, MD, MS, Frank M. Calia, MD Endowed Professor and Interim Chief, Division of Geographic Medicine, Department of Medicine (Sponsor Representative), University of Maryland, Baltimore
Organization: University of Maryland, Baltimore (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DMID 23-0015
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-05

CONDITIONS: Lassa Fever
Keywords: Lassa
MeSH Terms: conditions — Lassa Fever | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: This is a phase 1, randomized, controlled, recipient- and observer-blinded, dose-escalation clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - LASSARAB+ aPHAD-SE Vaccine at 700rU or Active Comparator (AC) (Experimental): 4:1 randomization to investigational vaccine or active comparator (n=5)
  Interventions: Biological: LASSARAB+ aPHAD-SEat 700rU; Biological: HDCV Comparator
- Cohort 2 - LASSARAB+ aPHAD-SE Vaccine at 700rU or 1400rU or AC (Experimental): 11:4:3 randomization to investigational vaccine dose 700rU or 1400rU or active comparator (n=18)
  Interventions: Biological: LASSARAB+ aPHAD-SEat 700rU; Biological: HDCV Comparator; Biological: LASSARAB+ aPHAD-SEat 1400rU
- Cohort 3 - LASSARAB+ aPHAD-SE Vaccine at 1400rU Single or Double or AC or AC/Placebo (Experimental): 11:2:4:1 randomization to investigational vaccine single dose at 1400rU or investigational vaccine (2 doses) at 14rU or active comparator or active comparator and normal saline placebo
  Interventions: Biological: HDCV Comparator; Other: Normal Saline Placebo; Biological: LASSARAB+ aPHAD-SEat 1400rU
- Cohort 4 - LASSARAB+ aPHAD-SE Vaccine at 1400rU (single) or AC/Placebo (Experimental): 11:3 randomization to investigational vaccine (2 doses) at 14rU or active comparator and normal saline placebo
  Interventions: Biological: HDCV Comparator; Other: Normal Saline Placebo; Biological: LASSARAB+ aPHAD-SEat 1400rU

INTERVENTIONS:
Biological: LASSARAB+ aPHAD-SEat 700rU — Rabies-Vectored Monovalent Lassa Fever Vaccine (LASSARAB) with 3D-(6- acyl) Phosphorylated Hexaacyl Disaccharides (PHAD)-Stable squalene oil-in-water nanoemulsion (aPHAD-SE) adjuvant administered by IM injection
  Arms: Cohort 1 - LASSARAB+ aPHAD-SE Vaccine at 700rU or Active Comparator (AC); Cohort 2 - LASSARAB+ aPHAD-SE Vaccine at 700rU or 1400rU or AC
Biological: HDCV Comparator — Sterile, stable, freeze-dried suspension of rabies virus prepared from strain PM-1503-3M
  Other Names: Imovax
Other: Normal Saline Placebo — Sterile 0.9% sodium chloride for injection, USP, or normal saline, is a sterile, nonpyrogenic, isotonic solution; each mL contains sodium chloride 9 mg
  Arms: Cohort 3 - LASSARAB+ aPHAD-SE Vaccine at 1400rU Single or Double or AC or AC/Placebo; Cohort 4 - LASSARAB+ aPHAD-SE Vaccine at 1400rU (single) or AC/Placebo
Biological: LASSARAB+ aPHAD-SEat 1400rU — Rabies-Vectored Monovalent Lassa Fever Vaccine (LASSARAB) with 3D-(6- acyl) Phosphorylated Hexaacyl Disaccharides (PHAD)-Stable squalene oil-in-water nanoemulsion (aPHAD-SE) adjuvant administered by IM injection
  Arms: Cohort 2 - LASSARAB+ aPHAD-SE Vaccine at 700rU or 1400rU or AC; Cohort 3 - LASSARAB+ aPHAD-SE Vaccine at 1400rU Single or Double or AC or AC/Placebo; Cohort 4 - LASSARAB+ aPHAD-SE Vaccine at 1400rU (single) or AC/Placebo

SUMMARY:
This study proposes the evaluation of a novel, first-in-human Lassa fever vaccine based on the complete Lassa glycoprotein complex (GPC) antigen. The antigen will be presented on a genetically modified and attenuated rabies vector expressing both the rabies glycoprotein (GP) antigen and the Lassa GPC. The inactivated chimeric virus is delivered with a toll-like receptor (TLR-4)-activating oil-in-water emulsion adjuvant. Studies using this vaccine administered as a prime-boost series in mice and non-human primates, and then challenged with Lassa virus demonstrated significant protection against Lassa fever. Given that the vaccine backbone is an attenuated and inactivated rabies virus expressing rabies GP, this vaccine will also be evaluated for immunogenicity against rabies virus.

DETAILED DESCRIPTION:
Lassa fever is a zoonotic infection endemic in West Africa and is spread by the Lassa virus, an arenavirus causing hemorrhagic fever. Up to 300,000 Lassa fever infections occur annually and while disease is often mild, in a subset of individuals disease is characterized by severe anemia, bleeding, encephalopathy, respiratory failure, shock, and high mortality. In some regions of West Africa, up to 15% of hospital admissions are secondary to Lassa fever, and an estimated 5,000 deaths occur annually. During epidemics of disease, case-fatality rates may reach as high as 50% in hospitalized patients. Approximately one-third of infected individuals will develop hearing loss regardless of disease severity, and in a proportion of patients, permanent deafness occurs.

Prevention of illness through vaccination is a critical goal in reducing the burden of disease from Lassa fever. There are currently no vaccines or therapeutics demonstrated to be efficacious in the prevention or treatment of Lassa fever. This study proposes the evaluation of a novel, first-in-human Lassa fever vaccine based on the complete Lassa glycoprotein complex (GPC) antigen. The antigen will be presented on a genetically modified and attenuated rabies vector expressing both the rabies glycoprotein (GP) antigen and the Lassa GPC. The inactivated chimeric virus is delivered with a toll-like receptor (TLR-4)-activating oil-in-water emulsion adjuvant. Studies using this vaccine administered as a prime-boost series in mice and non-human primates, and then challenged with Lassa virus demonstrated significant protection against Lassa fever. Given that the vaccine backbone is an attenuated and inactivated rabies virus expressing rabies GP, this vaccine will also be evaluated for immunogenicity against rabies virus.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to the initiation of any trial procedures.
2. Able to understand and agrees to comply with all planned trial procedures and be available for all study visits.
3. Age ≥ 18 and ≤50 years at time of enrollment.
4. In good general health and without clinically significant medical, psychiatric, chronic or intermittent health conditions including those listed in Exclusion Criteria
5. Participants of childbearing potential must have a negative serum human chronic gonadotropin (HCG) pregnancy test at screening and a negative urine HCG pregnancy test within 24 hours prior to the study vaccination.
6. Participants of childbearing potential in a heterosexual relationship agree to use of highly effective contraception beginning at the time of the screening visit through Day 61 (32 days after the last study treatment).
7. Vital signs and Body Mass Index (BMI) are in the following ranges at screening:

   * Oral temperature is less than 100.4°F (38.0°C).
   * Pulse is 47 to 100 beats per minute, inclusive.
   * Systolic blood pressure (SBP) is 85 to 140 mmHg, inclusive.
   * Diastolic blood pressure(DBP) is 55 to 90 mmHg, inclusive.
   * BMI of 18 kilograms/square meter (kg/m2) (inclusive) to <35 kg/m2
8. Has a negative test result for hepatitis B virus (HBV) surface antigen, hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening.
9. Has a negative rabies neutralizing antibody test at screening (< 0.5 IU/mL in RFFIT assay)
10. Screening hematology tests (white blood cells, hemoglobin, and platelets) and screening chemistry tests (alanine transaminase, creatine, and total bilirubin) are within acceptable parameters
11. Must agree to the collection and storage of residual biological specimens and additional clinical specimens for secondary research use
12. Agreement to adhere to Lifestyle Considerations during the study

Exclusion Criteria:

1. A history of anaphylaxis, serum sickness, meningitis; neuroparalytic events such as encephalitis, transient paralysis; Guillain-Barré Syndrome; myelitis; retrobulbar neuritis; history of prior or current hearing loss as assessed by quantitative audiometry; or multiple sclerosis
2. Current use of any medications that may be associated with impaired immune responsiveness
3. Allergy treatment with antigen injections within 60 days before first vaccination or that are planned through the end of the study.
4. Receipt of immunoglobulins and/or any blood products within the 60 days before first vaccination or that are planned through the end of the study.
5. Current pregnancy or lactation
6. Known allergic reactions to 1) any rabies vaccine; 2) any components of HDCV (human albumin, neomycin sulfate, phenol red, beta-propiolactone); 3) any components of LASSARAB +aPHAD-SE (LASSARAB, Tris-HCI, L-Arginine, (3D -(6-Acyl) PHAD, Squalene Redistilled, DMPC, Vitamin E Dry Powder).
7. History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions to drug or vaccine products.
8. Has a significant acute illness (with or without fever), as determined by the site PI or appropriate sub-investigator, within 72 hours prior to enrollment
9. Receipt of a rabies vaccine or an antibody therapeutic product for treating rabies or a Lassa fever vaccine any time before the first planned study vaccination.
10. Receipt of another experimental agent or intervention within 60 days before first vaccination or plans to do so before the end of the study.
11. Received or plans to receive any other vaccine in the 2 weeks prior to the first vaccination through Day 61 (32 days after the last study treatment).
12. Received or plans to receive any live vaccine in the 4 weeks prior to first vaccination through Day 61 (32 days after the last study treatment).
13. Self-reported or known history of alcoholism within the last 2 years.
14. Any condition that, in the judgment of the investigator, precludes participation because it could affect participant safety or endpoint assessment.
15. Has tattoos, scars, or other marks which would, in the opinion of the investigator, interfere with assessment of the vaccination site.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing solicited local and systemic events | From Day 1 through Day 8 for the first vaccination and from Day 29 through Day 36 for the second vaccination, as applicable
  Number of participants experiencing solicited local and systemic reactogenicity Adverse Events (AEs)
Percentage of participants experiencing solicited local and systemic events | From Day 1 through Day 8 for the first vaccination and from Day 29 through Day 36 for the second vaccination, as applicable
  Percentage of participants experiencing solicited local and systemic reactogenicity Adverse Events (AEs)
Number of participants experiencing unsolicited events | Day 1 through Day 61
  Number of participants experiencing any unsolicited AEs
Percentage of participants experiencing unsolicited events | Day 1 through Day 61
  Percentage of participants experiencing any unsolicited AEs
Number of participants experiencing Serious Adverse Events (SAEs) | Day 1 through Day 394
  Number of participants experiencing SAEs
Percentage of participants experiencing Serious Adverse Events (SAEs) | Day 1 through Day 394
  Percentage of participants experiencing SAEs
Number of participants experiencing Medically-Attended Adverse Events (MAAEs) | Day 1 through Day 394
  Number of participants experiencing MAAEs
Percentage of participants experiencing Medically-Attended Adverse Events (MAAEs) | Day 1 through Day 394
  Percentage of participants experiencing MAAEs
Number of participants experiencing New-Onset Chronic Medical Conditions (NOCMCs) | Day 1 through Day 394
  Number of participants experiencing NOCMCs
Percentage of participants experiencing New-Onset Chronic Medical Conditions (NOCMCs) | Day 1 through Day 394
  Percentage of participants experiencing NOCMCs
Number of participants experiencing Potential Immune-Mediated Medical Conditions (PIMMCs) | Day 1 through Day 394
  Number of participants experiencing PIMMCs
Percentage of participants experiencing Potential Immune-Mediated Medical Conditions (PIMMCs) | Day 1 through Day 394
  Percentage of participants experiencing PIMMCs
Number of participants experiencing Adverse Event of Special Interest (AESI) | Day 1 through Day 394
  Number of participants experiencing Adverse Event of Special Interest (AESI) - new onset sensorineural hearing loss (SNHL)
Percentage of participants experiencing Adverse Event of Special Interest (AESI) | Day 1 through Day 394
  Percentage of participants experiencing Adverse Event of Special Interest (AESI) - new onset sensorineural hearing loss (SNHL)
Number of participants experiencing clinical laboratory AEs | Day 1 through Day 61
  Number of participants experiencing clinical laboratory AEs
Percentage of participants experiencing clinical laboratory AEs | Day 1 through Day 61
  Percentage of participants experiencing clinical laboratory AEs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, University of Maryland School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States